CLINICAL TRIAL: NCT05646576
Title: Defining the Role of Palliative carE for Patients With Hematologic Malignancies Undergoing Adoptive CEllular Therapy: The PEACE Study
Brief Title: Defining the Role of Palliative carE for Patients With Hematologic Malignancies Undergoing Adoptive CEllular Therapy
Acronym: PEACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Principal Investigator, Patrick C. Johnson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-487
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hematologic Malignancy; Blood Cancer; Lymphoma; Leukemia; Multiple Myeloma
Keywords: Hematologic Malignancy; Adoptive Cellular Therapy; Palliative Care Intervention; Lymphoma; Leukemia; Multiple Myeloma; Palliative Care
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Leukemia; Multiple Myeloma | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care Intervention (PEACE) Group (Experimental): Participants will be randomly assigned, and stratified by disease, to the PEACE Group.
  * Participants will meet with palliative care (PC) clinician within 1 week of T-cell collection and within 72 hours of hospital admission for ACT.
  * Participants will meet with PC clinician at least 2 x weekly during hospitalization.
  * PC clinician will follow participants up to one year after randomization (or enrollment for the open pilot) and will meet participant at least 2 x weekly during inpatient hospitalizations.
  * Participants will complete follow-up study assessments on pre-determined days per protocol. The assessments will be filled out remotely or via paper.
  * Participants will complete exit interviews in the open pilot only.
  Interventions: Behavioral: Palliative Care
- Usual Care Group (Active Comparator): Participants will be randomly assigned, and stratified by disease, to the Usual Care Group and will receive standard care for ACT.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Palliative Care — * Palliative care (PC) intervention tailored to ACT recipients and addressing multiple PC domains with the input of ACT clinical experts, PC clinicians, and patients and caregivers.
  * Domains discussed include therapeutic relationship, symptom management, prognostic awareness and illness understanding, coping with illness, treatment decision-making, EOL care.
  * The palliative care intervention will be refined for the randomized control trial based on the feedback from the open pilot.
  Other Names: PEACE
  Arms: Palliative Care Intervention (PEACE) Group
Behavioral: Usual Care — Standard care for ACT per the treating team.
  Arms: Usual Care Group

SUMMARY:
The goal of this study is to determine whether a palliative care intervention (PEACE) can improve the quality of life and experiences of participants with Lymphoma, Leukemia, or Multiple Myeloma receiving adoptive cellular therapy (ACT). After completion of an open pilot, participants will be randomly assigned into one of two study intervention groups.

The names of the study intervention groups involved in this study are:

* Palliative care (PEACE) plus usual oncology care
* Usual care (standard oncology care)

Participation in this research study is expected to last for up to 2 years.

It is expected that about 90 people will take part in this research study.

DETAILED DESCRIPTION:
This is a single-center, parallel-group, randomized controlled study to determine whether a palliative care intervention (PEACE) can improve the quality of life and experiences of participants with Lymphoma, Leukemia, or Multiple Myeloma receiving adoptive cellular therapy (ACT).

10 participants with planned ACT will be enrolled into an open pilot and will receive a palliative care intervention (PEACE) for the duration of treatment. Once the palliative care intervention has been refined by feedback from the pilot participants, the study will enroll 80 participants and will randomly assign the participants into one of two study intervention groups. Randomization means that a participant is put into a group by chance.

The names of the study intervention groups involved in this study are:

* Palliative care intervention (PEACE) plus usual oncology care
* Usual care (standard oncology care)

Participation in this research study is expected to last for up to 2 years.

It is expected that about 90 people will take part in this research study.

The American Society of Clinical Oncology is supporting this research study by providing funding support.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Ability to complete surveys in English or with assistance of an interpreter.
* Diagnosis of a hematologic malignancy.
* Receiving autologous adoptive cellular therapy (ACT) at MGH with an FDA approved cellular therapy product.

Exclusion Criteria:

* Impaired cognition or uncontrolled mental illness that prohibits study compliance based on the oncology clinician assessment.
* Already receiving palliative care (PC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Eligible Participants Enrolled to Palliative Care Intervention (PEACE) (Feasibility) | 1 day
  Defined as at least 60% of eligible participants enrolling in the study, and among those enrolled and randomized to PEACE, 80% receiving PEACE as intended.

SECONDARY OUTCOMES:
Acceptability | Up to Day 90
  Defined as at least 80% of participants reporting satisfaction with PEACE on an adapted version of the Client Satisfaction Questionnaire with scores >=20.
Quality of Life - FACT-G | Baseline to day 90
  Defined by Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item questionnaire that assesses cancer domains of physical well-being, social/family well-being, and emotional and functional well-being.
Anxiety Symptoms | Baseline to day 90
  Assessed by the self-reported Hospital Anxiety and Depression Scale (HADS), which is a 14-item measure with subscales to evaluate symptoms of anxiety and depression. The HADS consists of two subscales assessing depression and anxiety symptoms, with scores ranging from 0 (no distress) to 21 (maximum distress)
Depression Symptoms | Baseline to day 90
  Assessed by the self-reported Hospital Anxiety and Depression Scale (HADS), which is a 14-item measure with subscales to evaluate symptoms of anxiety and depression. The HADS consists of two subscales assessing depression and anxiety symptoms, with scores ranging from 0 (no distress) to 21 (maximum distress)
Post-Traumatic Stress Disorder (PTSD) Symptoms | Baseline to day 90
  Defined by Post-Traumatic Stress Disorder Checklist (PCL), comprised of 17 items that corresponds to key symptoms of PTSD.
Physical Symptom Burden | Baseline to day 90
  Defined by Edmonton Symptom Assessment (ESAS-R), which is a 10-item measure to assess symptoms relevant to patients undergoing adoptive cellular therapy
Coping | Baseline to day 90
  Defined by Brief COPE which is comprised of 14 items that assesses the degree to which a participant utilizes specific coping strategies.
Prognostic Understanding | Baseline to day 90
  Defined by Perception of Treatment and Prognosis (PTPQ), a survey that assesses participant understanding of illness and prognosis.
End-of-Life Communication | Baseline to day 90
  Defined by PTPQ, a survey that assesses participant understanding of illness and prognosis and includes an item on patient-reported end-of-life communication.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick C Johnson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation